CLINICAL TRIAL: NCT05066048
Title: Intestinal Microecological Dysregulation Caused by Appendectomy Increases the Risk of Colorectal Cancer
Acronym: IMDCBAITROCC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2020-004
Record Dates: First submitted 2021-04-07; First posted 2021-10-04 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The appendectomy group
- Colorectal cancer group
- Normal group

SUMMARY:
As a good niche for bacterial growth, appendix plays a very important role in maintaining and protecting intestinal symbiotic flora. Appendectomy will lead to intestinal microecological disorders. Therefore, we put forward the hypothesis that "appendectomy leads to intestinal microecological disorders and then increases the risk of colorectal cancer". In this study, the feces of normal controls, appendectomy and patients with colorectal cancer were collected, and the specific changes of intestinal flora after appendectomy were explored in detail from the level of family, genus and species by macrogenomic sequencing. Then through functional gene analysis, metabolic pathway analysis and other methods to explore the molecular mechanism of colorectal cancer risk changes and the changes of microflora involved, and verified by mouse fecal bacteria transplantation animal experiment.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing appendectomy due to appendicitis;
* 6-36 months after appendectomy;
* Patients with no obvious abnormality observed by colonoscopy;
* Age between 20 and 85.

Exclusion Criteria:

* A. Any history of malignancy or disease
* Any inflammatory bowel disease (IBD) prior to study inclusion;
* Antibiotics and hormone drugs taken within the last three months;
* Patients with severe systemic diseases (severe diabetes, hypertension or autoimmune diseases, etc.);
* Severe clinical symptoms of digestive tract (severe diarrhea, constipation, purulent disease, etc.) within half a year.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with an appendectomy and meet the above conditions
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Species composition of fecal microbial | 1 year
  The types of microorganisms of fecal microbial

SECONDARY OUTCOMES:
weight in kilograms | baseline, pre-procedure
  weight of enrolled patients
height in meters | baseline, pre-procedure
  height of enrolled patients
age in year | baseline, pre-procedure
  age of enrolled patients

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi, China